CLINICAL TRIAL: NCT04315103
Title: Efficacy of a Single Crosslinked Hyaluronan (HYAJOINT Plus) Combined With a Single Platelet-rich Plasma (PRP) Versus a Single PRP for the Treatment of Knee Osteoarthritis: A Randomized-Controlled Trial
Brief Title: a Single HYAJOINT Plus Combined With a Single PPR Versus a Single PRP for Knee OA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Shu-Fen Sun, Director or Neurorehabilitation, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS107-152
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Knee OA
Keywords: Hyaluronan; Knee osteoarthritis; Platelet-rich plasma
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Patients with symptomatic knee OA were randomized to receive a single intraarticular injection of HYAJOINT Plus (3 ml) followed by 3 ml PRP (the combined-injection group) or a single injection of 3 ml PRP (the one-injection group).
Who Masked: Outcomes Assessor
Masking Description: Study blinding was accomplished by having an investigator (blinded to the randomization and treatment) perform all the assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the combined-injection group (Experimental): patients received a single intraarticular injection of HYAJOINT Plus (3 ml) followed by 3 ml PRP
  Interventions: Combination Product: a single intraarticular injection of HYAJOINT Plus (3 ml) followed by 3 ml PRP
- the one-injection group (Active Comparator): patients received a single injection of 3 ml PRP
  Interventions: Combination Product: a single intraarticular injection of HYAJOINT Plus (3 ml) followed by 3 ml PRP

INTERVENTIONS:
Combination Product: a single intraarticular injection of HYAJOINT Plus (3 ml) followed by 3 ml PRP — All the injections were done by the same experienced physician using aseptic procedures.
  Other Names: the one-injection group received a single injection of 3 ml PRP

SUMMARY:
Intraarticular hyaluronan or platelet-rich plasma (PRP) is each effective in the treatment for knee osteoarthritis (OA). The efficacy of combined hyaluronan with PRP for knee OA remained unclear. This study aimed to investigate the efficacy of a single intraarticular hyaluronan (HYAJOINT Plus) combined with a single PRP versus a single intraarticular PRP in patients with knee OA.

DETAILED DESCRIPTION:
Intraarticular HA or PRP has been used for knee OA for years. Combined HA and PRP has not been widely used for OA because of lack of clinical evidence. Based on in vitro and animal studies, combining HA and PRP may benefit from their dissimilar biological mechanisms for tissue repair and have potentials to synergistically promote cartilage regeneration, inhibit OA inflammation, modulate the disease process, and improve joint homeostasis in OA. Combination of HA and PRP has much potential for the treatment of OA, but the clinical evidence of this combination remains unclear. The purpose of this study was to investigate the efficacy and safety of combined a single crosslinked HA (HYAJOINT Plus) with a single PRP versus a single PRP alone in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-75 years;Symptomatic knee OA > 6 months despite conservative treatment such as oral analgesics, NSAIDs and/or physical therapy;Kellgren-Lawrence grades 2 knee OA on radiographs taken within the previous 6 months;Average pain at walking > 30 mm on a 100-mm visual analog scale (VAS);Radiological evidence of bilateral knee OA was accepted if global pain VAS in the contralateral knee< 30 mm.

Exclusion Criteria:

* Previous orthopedic surgery on the spine or lower limbs Disabling OA of either hip or foot Knee instability, apparent joint effusion or marked valgus/varus deformity Known allergy to hyaluronan products Women ascertained or suspected pregnancy or lactating Intraarticular injections into the knee in the past 6 months Any specific medical conditions (rheumatoid arthritis, active infections, severe cardiovascular diseases, autoimmune diseases, hemiparesis, neoplasm, etc.) that would interfere with the assessments

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
VAS pain score change from baseline | 1,3 and 6 months
  . The patient rated the average severity of knee pain on knee movement over the previous week on a 0-100 mm VAS (0=no pain to 100=worst possible pain)

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC, Likert Scale) | 1,3 and 6 months
  a 24-item questionnaire with 3 subscales measuring pain, stiffness, and physical function. Total score is 96 and higher scores indicate worse outcomes.
Lequesne index | 1,3 and 6 months
  used to assess severity of knee symptoms during the last week. It includes the measurement of pain, walking distance, and activities of daily living. Maximal score is 24 and higher scores represent worse function.
Single-leg stance test (SLS) | 1,3 and 6 months
  done by raising one foot up without touching it to the supported lower extremity with target knee and maintain balance for as long as possible. Each participant performed 3 trials, and the best result of the 3 trials was recorded.
satisfaction | 1,3 and 6 months
  Patients were asked to rate their treatment satisfaction compared to the preinjection condition, using a 100 mm VAS (0= completely dissatisfied, 100=completely satisfied).
consumption of analgesics | 1,3 and 6 months
  Acetaminophen (500mg; maximum daily dose, 4 g) was the only rescue medication allowed for knee pain. Acetaminophen was not permitted during the 24-hour period prior to each study visit. Use of rescue medication during the study period was recorded in a patient diary.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Fen Sun, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (2):
- Taiwan (2):
  - Department of Physical Medicine and Rehabilitation, Veterans General Hospital,, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun SF, Lin GC, Hsu CW, Lin HS, Liou IS, Wu SY. Comparing efficacy of intraarticular single crosslinked Hyaluronan (HYAJOINT Plus) and platelet-rich plasma (PRP) versus PRP alone for treating knee osteoarthritis. Sci Rep. 2021 Jan 8;11(1):140. doi: 10.1038/s41598-020-80333-x. PMID 33420185